CLINICAL TRIAL: NCT02727946
Title: Central Venous-arterial Carbon Dioxide Pressure Difference in Correlation to Dynamic Changes of Serum Lactate as an Indicator of Tissue Perfusion in Polytruama Patients
Brief Title: Tissue Perfusion Indices as Predictor of Outcome in Poly Trauma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Lecturer of Anesthesia and critical care Medicine, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00009902
Record Dates: First submitted 2016-03-23; First posted 2016-04-05 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-04

CONDITIONS: Multiple Trauma
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- optimal resuscitation (Other): This group of multiple trauma patients will be resuscitated with crystalloids, analgesics, blood products as needed. Then follow up of the difference between arterial and venous CO2 to difference between arterial and venous oxygen tension, serum lactate, renal function, other organ affection along over the short hospital stay period
  Interventions: Other: optimal resuscitation

INTERVENTIONS:
Other: optimal resuscitation — optimal resuscitation to achieve mean arterial blood pressure above 65 mmHG , Central venous pressure more than 8 mmHg , urine out put more than 0.5 ml /Kg/hour

SUMMARY:
Early intervention and resuscitation based upon a lot of clinical, laboratory findings make a big difference regarding outcome in poly trauma patients, the study uses the dynamic lactate change and the difference between arterial and venous CO2, oxygen tension or content as indicators for tissue perfusion.

DETAILED DESCRIPTION:
Poly trauma patients have high incidence of mortality and morbidity in spite of improvements and advances in facilities. However, no doubt that early resuscitation and interventions make a big difference upon the overall outcome.

A lot of methods, indices, laboratory and biomarkers have been utilized to evaluate the progress and quality of resuscitation and the early hospital interventions in such group of critically ill patients including central venous pressures, urine output, mixed venous oxygen saturation, and gastric tonometry. Most of recent means focus upon the regional tissue perfusion rather than global, however some researches have tried the difference between arterial and venous CO2,oxygen tension or content ( Pv -a co2& Pa -v O2 ) in addition to dynamic changes in lactate(3) as predictors for tissue perfusion in sepsis patients after establishment of sepsis campaign (bundle).

ELIGIBILITY:
Inclusion Criteria:

* multiple trauma patients Adult patients

Exclusion Criteria:

* cardiac renal chronic chest disease diabetic more than 3 years

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-09 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
the difference between partial pressure of oxygen in arterial and venous blood | 6 hours
the difference between partial pressure of carbon dioxide in arterial and venous blood | 6 hours
serum level of lactate and its changes | 6 hours
  as an index for tissue oxygenation

SECONDARY OUTCOMES:
Kidney function | 72 hours
  serum creatinine in mg/ dl and urine output/ hour
hemodynamic stability including pulse rate and mean arterial blood pressure | 72 hours
duration of stay in the critical care unit | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Emad Zarief Kamel Said, MD, Study Director — Assiut University
Locations (1):
- Emad Zarief Kamel Said, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No